CLINICAL TRIAL: NCT07327190
Title: Effects of Motor Imagery and Action Observation Training on Pain, Functionality, Balance and Fear of Movement in Total Knee Arthroplasty: A Randomized Controlled Trial.
Brief Title: Motor Imagery and Action Observation Training in Total Knee Arthroplasty: A Randomized Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KSBU-TDA
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis; Knee Disease
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Traditional Physiotherapy) (Active Comparator): Standard physiotherapy exercise routines will include: ankle pumping exercises, passive/active/active assisted hip flexion (straight leg raise), abduction/adduction, passive/active/active assisted hip-knee flexion (starting from 30°-40°), isometric exercises (quadriceps, adductor, gluteal muscles, hamstrings), cryotherapy (3 times a day), and stretching exercises (hamstring, gastro-soleus), along with walker assistance for standing, walking training, and stair training. In addition, participants in this group will be given recordings containing nature sounds and nature videos to listen to and watch after their exercises.
  Interventions: Other: Traditional Physiotherapy
- Motor imagery group (Experimental): In motor imagery training, participants will visualize standard physiotherapy tasks using audio recordings presented as metaphors. Participants will be asked to fully focus on visualizing the movements in a quiet environment. They will also be asked to imagine different activities from daily life, progressing from simple to more challenging. Patients will undergo imagery training with audio recordings of standard physiotherapy exercises for six weeks. The training content will parallel the standard physiotherapy program. Participants in the motor imagery training group will be provided with audio explanations (mp3 files) of the motor imagery session instructions to continue at home. Patients in this group will also watch videos containing nature visuals.
  Interventions: Other: Motor imagery training
- Action observation group (Experimental): In the action observation group, participants will observe movements by watching videos of standard physiotherapy tasks in addition to standard physiotherapy. The training content will progress in parallel with the standard physiotherapy program. The training content will be prepared by clearly recording frontal or lateral views of all exercises included in the standard physiotherapy curriculum (0-2 week, 2-6 week exercises). Patients in this group will also listen to an audio recording containing relaxing music.
  Interventions: Other: Action observation training

INTERVENTIONS:
Other: Traditional Physiotherapy — Patients will be given a standard physiotherapy program consisting of 0-2 weeks and 2-6 weeks, with the first week mainly featuring isometric exercises, stretching exercises, and ankle pumping exercises, and the second-6 weeks transitioning to strengthening exercises.
  Arms: Control Group (Traditional Physiotherapy)
Other: Motor imagery training — In addition to standard visual therapy, patients will be sent audio recordings that allow them to visualize movement; they will also be sent nature videos.
  Arms: Motor imagery group
Other: Action observation training — In this group, in addition to standard physiotherapy, participants will be given videos showing visuals of the movements and will also be sent audio recordings containing nature sounds during the session.
  Arms: Action observation group

SUMMARY:
This single-center randomized controlled trial aims to evaluate the effects of motor imagery and action observation training on pain, functionality, balance, and fear of movement in patients after total knee arthroplasty (TKA). The study will be conducted at Simav Doç. Dr. İsmail Karakuyu State Hospital Orthopedics Department with a minimum of 40 participants meeting the inclusion criteria. Participants will be randomly assigned to one of three groups: (1) standard physiotherapy, (2) standard physiotherapy plus motor imagery training, or (3) standard physiotherapy plus action observation training.

All interventions will last six weeks. Standard physiotherapy will include ankle pumping, active-assisted hip and knee flexion, isometric and stretching exercises, cryotherapy, gait, and stair training. The motor imagery group will perform guided imagery sessions using audio recordings describing the physiotherapy exercises and daily activities. The action observation group will observe exercise videos corresponding to the physiotherapy program.

The primary outcomes will include pain, functional level, balance, and kinesiophobia. The study aims to determine whether the addition of mental simulation techniques to standard physiotherapy can enhance postoperative recovery and improve functional outcomes in patients undergoing total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Those diagnosed with degenerative gonarthrosis and who have experienced unilateral TDA
* Those over 25 years of age
* Those who have obtained a passing score on the Mini Mental Test (>24)

Exclusion Criteria:

* Body mass index of 40 kg/m2 or higher,
* Revision/bilateral TDA,
* Self-reported sensory, cognitive, neurological or motor impairment that would limit participation in the study; history of psychosis; or concomitant diseases that would negatively affect recovery, such as hemiparesis, peripheral neuropathy, lymphedema or lower extremity amputation.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2025-10-14 (Actual); Primary Completion 2026-03-03 (Estimated); Study Completion 2026-05-03 (Estimated)

PRIMARY OUTCOMES:
Pain Assessment | a day before the operation
  Pain intensity will be measured using a Visual Analog Scale.
Pain Assessment | after 2 weeks of operation
  Pain intensity will be measured using a Visual Analog Scale.
Pain Assessment | after 6 weeks of operation
  Pain intensity will be measured using a Visual Analog Scale.
Muscle Strength Assessment: | a day before the operation
  Muscle strength will be measured using a handheld dynamometer (Lafayette Instrument®) located in the physiotherapy unit, with the knee in a 90° flexion position. The device will be placed on the front surface above the malleoli of the ankle. A maximum isometric contraction in the extension direction will be requested against the device for 5 seconds. Three repetitions of the movement will be performed, and the average will be taken. A 30-second rest break will be given between each contraction. Measurements will be recorded in kilograms. The muscle strength measuring instrument will be obtained from the physiotherapy unit.
Muscle Strength Assessment: | after 2 weeks of operation
  Muscle strength will be measured using a handheld dynamometer (Lafayette Instrument®) located in the physiotherapy unit, with the knee in a 90° flexion position. The device will be placed on the front surface above the malleoli of the ankle. A maximum isometric contraction in the extension direction will be requested against the device for 5 seconds. Three repetitions of the movement will be performed, and the average will be taken. A 30-second rest break will be given between each contraction. Measurements will be recorded in kilograms. The muscle strength measuring instrument will be obtained from the physiotherapy unit.
Muscle Strength Assessment: | after 6 weeks of operation
  Muscle strength will be measured using a handheld dynamometer (Lafayette Instrument®) located in the physiotherapy unit, with the knee in a 90° flexion position. The device will be placed on the front surface above the malleoli of the ankle. A maximum isometric contraction in the extension direction will be requested against the device for 5 seconds. Three repetitions of the movement will be performed, and the average will be taken. A 30-second rest break will be given between each contraction. Measurements will be recorded in kilograms. The muscle strength measuring instrument will be obtained from the physiotherapy unit.
Functional Assessment | a day before the operation
  The WOMAC will be used for functional assessment. The WOMAC consists of sub-sections for pain, stiffness, and physical function. Higher scores indicate greater pain, stiffness, and worse physical function.
Functional Assessment | after 2 weeks of operation
  The WOMAC will be used for functional assessment. The WOMAC consists of sub-sections for pain, stiffness, and physical function. Higher scores indicate greater pain, stiffness, and worse physical function.
Functional Assessment | after 6 weeks of operation
  The WOMAC will be used for functional assessment. The WOMAC consists of sub-sections for pain, stiffness, and physical function. Higher scores indicate greater pain, stiffness, and worse physical function.
Timed Get Up and Walk (TUG) Test | a day before the operation
  This test will be used to assess physical performance. For the test, participants will be asked to get up from a seated position without holding onto the chair's arms, walk 3 meters, return to the chair, and walk back to sit down. The elapsed time will be measured and recorded using a stopwatch. The test will be repeated 3 times, and the average will be taken.
Timed Get Up and Walk (TUG) Test | after 2 weeks of operation
  This test will be used to assess physical performance. For the test, participants will be asked to get up from a seated position without holding onto the chair's arms, walk 3 meters, return to the chair, and walk back to sit down. The elapsed time will be measured and recorded using a stopwatch. The test will be repeated 3 times, and the average will be taken.
Timed Get Up and Walk (TUG) Test | after 6 weeks of operation
  This test will be used to assess physical performance. For the test, participants will be asked to get up from a seated position without holding onto the chair's arms, walk 3 meters, return to the chair, and walk back to sit down. The elapsed time will be measured and recorded using a stopwatch. The test will be repeated 3 times, and the average will be taken.
ROM Assessment | a day before the operation
  A standard goniometer will be used to assess active ROM. For knee flexion ROM, the fixed arm of the goniometer will be placed parallel to the long axis of the femur. The movable arm will be placed parallel to the long axis of the fibula. The participant will be asked to flex their knee without breaking contact between their foot and the bed. Extension angle will be measured using the same procedure after the heel is placed approximately 15 cm high and the participant is asked to perform active knee extension. Flexion and extension measurements will be repeated 3 times, and the averages will be recorded.
ROM Assessment | after 2 weeks of operation
  A standard goniometer will be used to assess active ROM. For knee flexion ROM, the fixed arm of the goniometer will be placed parallel to the long axis of the femur. The movable arm will be placed parallel to the long axis of the fibula. The participant will be asked to flex their knee without breaking contact between their foot and the bed. Extension angle will be measured using the same procedure after the heel is placed approximately 15 cm high and the participant is asked to perform active knee extension. Flexion and extension measurements will be repeated 3 times, and the averages will be recorded.
ROM Assessment | after 6 weeks of operation
  A standard goniometer will be used to assess active ROM. For knee flexion ROM, the fixed arm of the goniometer will be placed parallel to the long axis of the femur. The movable arm will be placed parallel to the long axis of the fibula. The participant will be asked to flex their knee without breaking contact between their foot and the bed. Extension angle will be measured using the same procedure after the heel is placed approximately 15 cm high and the participant is asked to perform active knee extension. Flexion and extension measurements will be repeated 3 times, and the averages will be recorded.
Assessment of Kinesiophobia | a day before the operation
  he Tampa Kinesiophobia Scale will be used. The Turkish validity and reliability of the TKÖ, a 17-question scale designed to measure fear of movement, was established by Tunca Yılmaz et al. in 2011. A 4-point Likert scale is used (Strongly disagree: 1, Disagree: 2, Agree: 3, Strongly agree: 4). Questions 4, 8, 12, and 16 are reverse Likert scales; the total scale score is calculated as 33. Individuals will receive a total score between 17 and 68. The higher the score on the scale, the higher the fear of movement.
Assessment of Kinesiophobia | after 2 weeks of operation
  he Tampa Kinesiophobia Scale will be used. The Turkish validity and reliability of the TKÖ, a 17-question scale designed to measure fear of movement, was established by Tunca Yılmaz et al. in 2011. A 4-point Likert scale is used (Strongly disagree: 1, Disagree: 2, Agree: 3, Strongly agree: 4). Questions 4, 8, 12, and 16 are reverse Likert scales; the total scale score is calculated as 33. Individuals will receive a total score between 17 and 68. The higher the score on the scale, the higher the fear of movement.
Assessment of Kinesiophobia | after 6 weeks of operation
  he Tampa Kinesiophobia Scale will be used. The Turkish validity and reliability of the TKÖ, a 17-question scale designed to measure fear of movement, was established by Tunca Yılmaz et al. in 2011. A 4-point Likert scale is used (Strongly disagree: 1, Disagree: 2, Agree: 3, Strongly agree: 4). Questions 4, 8, 12, and 16 are reverse Likert scales; the total scale score is calculated as 33. Individuals will receive a total score between 17 and 68. The higher the score on the scale, the higher the fear of movement.
The Standardized Mini Mental Test (SMMT) | a day before the operation
  It is a short, efficient, and standardized method that can be preferred for determining an individual's cognitive level. It is divided into five sections: orientation, recording memory, attention and calculation, recall, and language. There are eleven items for individuals to answer. It is evaluated out of a total of 30 points. The Turkish validity and reliability study was conducted by Güngen et al. In the validity and reliability study, the threshold value was determined as 24 points.
The Standardized Mini Mental Test (SMMT) | after 2 weeks of operation
  It is a short, efficient, and standardized method that can be preferred for determining an individual's cognitive level. It is divided into five sections: orientation, recording memory, attention and calculation, recall, and language. There are eleven items for individuals to answer. It is evaluated out of a total of 30 points. The Turkish validity and reliability study was conducted by Güngen et al. In the validity and reliability study, the threshold value was determined as 24 points.
The Standardized Mini Mental Test (SMMT) | after 6 weeks of operation
  It is a short, efficient, and standardized method that can be preferred for determining an individual's cognitive level. It is divided into five sections: orientation, recording memory, attention and calculation, recall, and language. There are eleven items for individuals to answer. It is evaluated out of a total of 30 points. The Turkish validity and reliability study was conducted by Güngen et al. In the validity and reliability study, the threshold value was determined as 24 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Health Sciences University, Kütahya, Turkey (Türkiye)